CLINICAL TRIAL: NCT06280170
Title: AI for All: Harnessing the Power of Artificial Intelligence in Mental Health Case Management
Brief Title: AI to Support Mental Health Case Management Providers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eleos Health (Industry)
Collaborators: Centerstone Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ST11480
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Depressive Disorder; Anxiety Disorders; Substance Use Disorders; Post Traumatic Stress Disorder
Keywords: Case management; Artificial Intelligence; Provider productivity; Mental health services; Provider satisfaction
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Substance-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Case Managers

STUDY DESIGN:
Intervention Model Description: This study will follow a stepped-wedge, randomized controlled design, where each provider team will undergo two phases: SAU and the AI platform phase. All teams will initially start with SAU, and the AI platform will be sequentially introduced to teams over time. Teams will be randomly assigned to different time periods for the AI platform phase using simple randomization. The order of implementation will be determined by randomly selecting the number of the team from sealed envelopes every two months. In both phases, the study will enroll new and existing clients. At the end of the trial all teams would have used Eleos for a few months
Masking Description: The masking in this study involves a differential approach between providers and clients. Providers will be aware of whether they are in the Services-As-Usual (SAU) or Artificial Intelligence (AI) phase. However, participating clients will not be informed about the platform their provider is using to document their therapy sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services-as-usual (SAU) (No Intervention): During the services-as-usual (SAU) phase of this study, providers will deliver the routine case management services offered by Centerstone and report these services in the usual way they do.
- Artificial Intelligence (AI) (Experimental): Once randomized to start using the AI-based platform for documenting their services, providers will have access to the Eleos Health platform, a secure and HIPAA-compliant tool specifically designed for documenting behavioral health encounters. This AI-powered platform enables providers to complete progress notes more quickly. Providers will complete the progress notes on their phones, and these notes will be integrated into the client's electronic health records.
  Interventions: Other: Artificial Intelligence platform for case managers

INTERVENTIONS:
Other: Artificial Intelligence platform for case managers — Providers will have access to the Eleos Health mobile AI platform to document their case management encounters.
  Arms: Artificial Intelligence (AI)

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of an artificial intelligence (AI) platform for case managers in a nonprofit health system specializing in mental health and substance use disorder. The main questions it aims to answer are:

1. Is the AI platform acceptable and feasible for case managers?
2. Does the AI platform improve providers' productivity and reported interventions? Participants will be approximately 30 case managers and their 250 adult clients receiving case management services. Researchers will compare the provider productivity and work satisfaction prior to the implementation of the AI platform to following its implementation.

ELIGIBILITY:
FOR PROVIDERS:

Participating providers must be Centerstone case managers.

FOR CLIENTS:

Inclusion Criteria:

1. Participants must be adults.
2. Participants must be receiving case management services from a Centerstone provider

Exclusion Criteria:

1. Participants currently involved in any other concurrent research study will be excluded to avoid potential confounding factors.
2. Participants with any medical conditions or medications that may significantly interfere with the study outcomes will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Case manager satisfaction | Baseline, and 4 months after the rollout of the Eleos Health tool.
  Providers will complete a self-report assessment about their experience providing case management services. Providers will be asked to (a) report the number of of hours spent on documentation per week; (b) respond on a Likert Scale (1-5, 1="Not at all" and 5="highly stressed" regarding their stress level about documentation; and (c) respond on a Likert scale 1-5 (1="Not at all satisfied", 5="Highly satisfied"), indicating their satisfaction with their current role as a case manager.
Case manager productivity | 3 months before and 3 month after study start date
  We will collect the number of encounters (i.e., case management visits provided) per month in the three months preceding the start of the study, and months 3-6 after the AI platform rollout.
Case manager note completion time | 3 months before and 3 month after study start date
  We will record progress note completion time by hours since the time of service delivery (average, standard deviation, and range).

SECONDARY OUTCOMES:
Clients' crisis services utilization | 6 months before and 6 month after study start date
  Data on the clients' healthcare crisis encounters reported in the system will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Centerstone, Alton, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The confidentiality and privacy of the participants' data are paramount, and sharing individual-level data could compromise their privacy. Therefore, the study does not include provisions for sharing IPD with other researchers.

REFERENCES:
- [Background] Kellogg KC, Sadeh-Sharvit S. Pragmatic AI-augmentation in mental healthcare: Key technologies, potential benefits, and real-world challenges and solutions for frontline clinicians. Front Psychiatry. 2022 Sep 6;13:990370. doi: 10.3389/fpsyt.2022.990370. eCollection 2022. PMID 36147984
- [Background] Sadeh-Sharvit S, Hollon SD. Leveraging the Power of Nondisruptive Technologies to Optimize Mental Health Treatment: Case Study. JMIR Ment Health. 2020 Nov 26;7(11):e20646. doi: 10.2196/20646. PMID 33242025
- [Background] Sadeh-Sharvit S, Camp TD, Horton SE, Hefner JD, Berry JM, Grossman E, Hollon SD. Effects of an Artificial Intelligence Platform for Behavioral Interventions on Depression and Anxiety Symptoms: Randomized Clinical Trial. J Med Internet Res. 2023 Jul 10;25:e46781. doi: 10.2196/46781. PMID 37428547
- See also: Link to Eleos Health's science page — https://eleos.health/science/
- See also: Link to Centerstone Research Institute — https://centerstone.org/locations/institute/